CLINICAL TRIAL: NCT07153172
Title: Safety Follow-up Study of Participants Previously Dosed With INV-347 in the First-in-Human Study INV-CL-108
Brief Title: Safety Follow-up Study of Participants Dosed With INV-347 in Study INV-CL-108
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NN9441-8452; U1111-1319-3945 (Other: WHO)
Record Dates: First submitted 2025-07-28; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants from the study INV-CL-108 (Experimental): Participants who were dosed with INV-347 in the First In Human study INV-CL-108 and still have measurable plasma exposure of INV-347 are included to assess long term safety.
  Interventions: Drug: INV-347

INTERVENTIONS:
Drug: INV-347 — Participants who were dosed with INV-347 in the First In Human study INV-CL-108 and still have measurable plasma exposure of INV-347 are included to assess long term safety.

SUMMARY:
The study looks at the safety and blood levels of the study drug INV-347 in participants who were previously dosed with INV-347 in study INV-CL-108. Participants will not get any study drug in this study as it looks into the safety of a drug previously dosed. The study will last for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female (sex at birth).
3. Age 18 years or above at the time of signing the informed consent.
4. Previously dosed with INV-347 in study INV-CL-108 and with measurable INV-347 concentration in plasma at enrolment [above lower limit of qualification (LLOQ) of 0.5 nanogram per milliliter (ng/mL)].

Exclusion Criteria:

The study has no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | From the end-of-study participation in INV-CL-108 (week 0) to completion of the end-of-study visit (up to week 104 from enrolment)
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Syneos Health, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com